CLINICAL TRIAL: NCT00196001
Title: G Protein Expression in Response to ACTH Stimulation Testing
Brief Title: Adrenocorticotropic Hormone (ACTH) Stimulation and G Protein
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 01.4204
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Adrenal Sufficiency
Keywords: Adrenal sufficiency; Low-dose ACTH stimulation; G proteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Males and females may exhibit different responses to testing of adrenal function. The hormones responsible for controlling adrenal function are ACTH (adrenocorticotropic hormone or corticotropin) and CRH (corticotropin-releasing hormone). Adrenal function is tested with an ACTH stimulation test. ACTH stimulates the adrenal glands to produce cortisol. Cortisol levels are measured, and a certain peak level indicates normal adrenal gland function. Females may produce more cortisol in response to ACTH testing than males. This difference may be due to certain proteins, called G proteins. The hormones controlling adrenal function, ACTH and CRH, work through G proteins. Females may have more G proteins than males allowing for the increased cortisol response to ACTH stimulation.

The investigators speculate that:

1. There may be differences in adrenal responsiveness to ACTH stimulation testing between healthy males and females.
2. ACTH and CRH induce their own function.
3. Sex differences in adrenal responsiveness to ACTH stimulation testing may be related to sex differences in G protein expression.

In this study, cortisol, a hormone produced by the adrenal glands, will be measured before and after the administration of ACTH.

This study will also measure G proteins. G proteins are found in the white blood cells. White blood cells from females may have more active G proteins than white blood cells from males. Sex differences may be augmented after exposure to ACTH.

DETAILED DESCRIPTION:
Many nonsteroidal hormones work through G protein signal transducers. These heterotrimeric signal transducers couple cell surface receptors to intracellular pathways, thus conveying biologic effects. Most hormones that work via the stimulatory G protein, Gas, also exert actions through a homologous stimulatory G protein, Gaq, suggesting that these pathways exhibit redundancy. We have previously demonstrated sex differences in the expression of Gas and Gaq. We have observed that female mice and humans display significantly higher levels of mRNA and protein for the G protein, Gaq. We have also observed that estrogens induce expression of Gaq mRNA and protein in female mice. In addition, preliminary studies in mice demonstrate that both ACTH (adrenocorticotropic hormone or corticotropin) and CRH (corticotropin-releasing hormone) induce Gaq in immune cells and adrenal tissue in a sex restricted fashion, i.e. females only.

ACTH and CRH are the two major hormones controlling adrenal function. Adrenal function can be tested using a standard 1mcg synthetic ACTH stimulation test and measuring the production of cortisol. We have observed that females exhibit a trend toward increased responsiveness to ACTH stimulation than males. We speculate that sex differences in cortisol responsiveness to ACTH exist, and that these differences will correlate with sex differences in the expression or induction of the G proteins, Gaq or Gas.

We propose to determine whether healthy female subjects undergoing low-dose ACTH stimulation exhibit altered levels of Gaq or Gas mRNA and protein and cortisol levels compared with male subjects undergoing the same provocative testing. This study may have implications for the interpretation of provocative ACTH testing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 6-60

Exclusion Criteria:

* Known medical condition
* Use of inhaled, topical, or oral steroids
* Use of oral contraceptive pills or hormone replacement
* Menopause
* Pregnancy

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy male and female subjects (ages 6-34)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill D Jacobson, MD, Study Director — Children's Mercy Hospital Kansas City; Kelly J Seiler, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Wayne V Moore, MD, PhD, Study Chair — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Morton TL, Ansari MA, Jacobson JD. Gender differences and hormonal modulation of G proteins Gaq/11 expression in lymphoid organs. Neuroendocrinology 2003;78:147-153. Clark PM, Neylon I, Raggatt PR, Sheppard MC, Stewart PM. Defining the normal cortisol response to the short Synacthen test: implications for the investigation of hypothalamic-pituitary disorders. Clin Endocrinol 1998;49:287-292. Dickstein G, Shechner C, Nicholson WE, Rosner I, Shen-Orr, Adawi F, et al. Adrenocorticotropin stimulation test: effects of basal cortisol level, time of day, and suggested new sensitive low dose test. J Clin Endocrinol Metab 1991;72:773-778. Tordjman K, Jaffe A, Grazas N, Apter C, Stern N. The role of the low dose (1 mcg) adrenocorticotropin test in the evaluation of patients with pituitary disease. J Clin Endocrinol Metab 1995;80:1301-1305. Thaler LM, Blevins LS. The low dose (1-mcg) adrenocorticotropin stimulation test in the evaluation of patients with suspected central adrenal insufficiency. J Clin Endocrinol Metab 1998;83:2726-2729. Dorin RI, Qualls CR, Crapo LM. Diagnosis of adrenal insufficiency. Ann Intern Med 2003;139:194-204. Product Information: Acthar(R), corticotropin. Armour Pharmaceutical, Blue Bell, PA, 1990. Jacobson JD, Ansari MA, Kinealy M, Muthukrishnan V. Gender-specific exacerbation of murine lupus by gonadotropin-releasing hormone: potential role of Gaq/11. Endocrinology 1999;140:3429-3437. Chomczynski P. A reagent for the single-step simultaneous isolation of RNA, DNA and proteins from cell and tissue samples. Biotechniques 1993;15(3):532-4, 536-7.